CLINICAL TRIAL: NCT04593979
Title: Virological Failure and HIV Drug Resistance Among Adolescents Receiving Antiretroviral Treatment in Cameroon
Brief Title: ANRS 12406 EvvA Study
Acronym: EvvA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Hospital Laquinitinie de Douala (Unknown); Franceville International Center for Medical Research, Gabon (Unknown); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: ANRS 12406 EvvA
Record Dates: First submitted 2020-10-05; First posted 2020-10-20 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: HIV-1-infection
Keywords: Virological failure; HIV drug resistance; Adolescents; Cameroon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ANRS 12406 EvvA is an observational, longitudinal and monocentric study evaluating the virological success rate in HIV-infected adolescents on antiretroviral therapy in Cameroon.

The main objective of the study is to estimate the rate of virological suppression among adolescents on antiretroviral therapy for more than 6 months in Cameroon

DETAILED DESCRIPTION:
At the end of 2017, HIV-AIDS affects more than 36 million people worldwide, more than three-quarters of whom live in sub-Saharan Africa, and a quarter of the infections are among young people and adolescents. Every hour, 4 adolescents (aged 15-19) are newly infected with HIV in the world, and 3 of them are adolescents. Three infections occur in sub-Saharan Africa, and for five adolescents living with HIV, there are seven girls (aged 10 to 19) in the same situation. This gender disparity increases when adolescents reach adulthood. This group of the population may well deserve the term "key and vulnerable population". In the era of international commitment to end the AIDS epidemic by 2030, especially to stop new infections, it is essential not to neglect part of the epidemic because it would effectively represent a reservoir for maintaining the epidemic and make these eradication goals impracticable. Data on virological success among adolescents on antiretroviral treatment are generally scarce and this is much more striking in Central Africa. Also, information on the frequency of emergence of resistant viruses and the consequences for the effectiveness of available treatments is rare. However, in the absence of such data, it is difficult, if not impossible, to take the right decisions to improve the care and monitoring of adolescents. In addition, the few available data indicate high virological failure rates and high frequencies of drug resistance, which may indicate a need to further investigate virological failure events in this population.

This study will be conducted in Cameroon among 289 adolescents during 9 months, where access to biological monitoring is a major challenge, especially with low access to viral load testing. The results of this project will inform on the current state of success of ARV treatments in this population. Moreover, the other goal of this study is to conclude on the need to conduct a larger study at the national or regional level according to the results obtained

ELIGIBILITY:
Inclusion Criteria:

* Being adolescent (aged 10 to 19) on antiretroviral therapy and followed at the Laquintinie Hospital (Douala Cameroon)
* HIV-1 infection
* Duration of antiretroviral therapy ≥ 6 months regardless of antiretroviral regimen
* For emancipated adolescents: obtaining informed consent signed by the adolescent
* For unemancipated adolescents:
* Obtaining informed consent signed by the legal representative (parent(s) or guardian(s))
* Obtaining the assent of adolescents able to understand the study (maturity and knowledge of HIV status)

Exclusion Criteria:

* Infection with HIV-1 or HIV-1/HIV2 co-infection

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include adolescents living with HIV infection, aged 10 to 19 years and follow-up in a treatment unit in Douala, Cameroon.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-01-14 (Estimated); Study Completion 2022-01-14 (Estimated)

PRIMARY OUTCOMES:
Viral load suppression after ≥ 6 months of antiretroviral therapy | Day 0
  Proportion of participants with HIV-1 RNA <1000 copies / ml after ≥ 6 months of antiretroviral therapy

SECONDARY OUTCOMES:
Drug resistance after ≥ 6 months of antiretroviral therapy | 3 months
  Proportion of participants with HIV-1 RNA ≥ 300 copies / ml and presence of antiretroviral-resistant virus (ARV) after ≥ 6 months of antiretroviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Avelin F AGHOKENG, PhD, Study Director — Institut de Recherche pour le Developpement; Ida C PENDA, Principal Investigator — Hôpital Laquinitie de Douala
Locations (1):
- Hôpital Laquinitie de Douala, Douala, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided
To be decided later

REFERENCES:
- [Derived] Djiyou ABD, Penda CI, Madec Y, Ngondi GD, Moukoko A, Varloteaux M, de Monteynard LA, Moins C, Moukoko CEE, Aghokeng AF. Viral load suppression in HIV-infected adolescents in cameroon: towards achieving the UNAIDS 95% viral suppression target. BMC Pediatr. 2023 Mar 15;23(1):119. doi: 10.1186/s12887-023-03943-0. PMID 36922769